CLINICAL TRIAL: NCT04478981
Title: The Natural History of Patients With Congenital Muscular Dystrophies Due to Mutations in the SELENON or LAMA2 Genes: Working Towards Trial-readiness in Two Mitochondrial Myopathy Mimics
Brief Title: The Natural History of Patients With Mutations in SEPN1 (SELENON) or LAMA2
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: NL64269.091.17
Record Dates: First submitted 2020-07-09; First posted 2020-07-21 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2022-04

CONDITIONS: MDC1A; SELENON-related Myopathy
Keywords: MDC1A; LAMA2-related muscular dystrophy; LAMA2; Laminin2 / genetics; Laminin2 / deficiency; SELENON; SEPN1; Multi-minicore Disease; Rigid Spine Muscular Dystrophy; Selenoproteins / genetics; Natural history study; Outcome measures; Congenital muscular dystrophy; Congenital myopathy; Muscle disease
MeSH Terms: conditions — Muscular dystrophy congenital, merosin negative; Rigid spine syndrome; Minicore Myopathy with External Ophthalmoplegia; Myotonia Congenita; Muscular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SELENON- or LAMA2-related muscular dystrophy: Participants diagnosed with congenital myopathy/muscular dystrophy due to mutations in the SEPN1 (SELENON) or LAMA2 gene
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — This concerns a natural history study; no interventions will be used

SUMMARY:
SEPN1 (SELENON) is a rare congenital myopathy due to mutations in the SELENON gene. MDC1A is a rare congenital muscle dystrophy due to mutations in the LAMA2 gene. Currently, not much is known about the natural history of these two muscle diseases and no (curative) treatment options exist. The investigators aim to study the natural history of SELENON- and LAMA2-related myopathy/congenital muscular dystrophy patients and prepare for future trials by selection of the most appropriate outcome measures. To this end, a standard medical history, neurological examination, functional measures, questionnaires, cardiac examination, respiratory function tests, radiological examination and accelerometry will be performed over an one and-a-half year period.

DETAILED DESCRIPTION:
Rationale: Patients with mutations in the SELENON gene suffer from slowly progressive congenital muscular dystrophy with early onset rigidity of the spine and potentially life-threatening respiratory insufficiency. The protein encoded by SELENON, selenoprotein-1, functions as an endogeneous antioxidant and executes a role in cellular redox metabolism. The first results of an intervention study using KH176, currently under development for mitochondrial disease, in an animal model (Sepn1 knock out zebrafish) showed improved muscular function. Patients with mutations in LAMA2 gene causing merosin-deficient congenital muscular dystrophy (MDC1A) have a similar phenotype as those with mutations in SELENON gene. Key characteristics include congenital hypotonia, delayed motor development and contractures. For them no treatment is available either. Since not much is known about the clinical progression of these two congenital muscle diseases, there is an urgent need for natural history-outcome measure studies to reach trial-readiness enabling smooth transition towards clinical trials.

Objective: The primary objective is to identify and follow (i.e. describe the natural history of) patients with congenital myopathy/muscular dystrophy due to mutations in SELENON- or LAMA2 genes. The secondary objectives are: 1. to select appropriate outcome measures based on the natural history data. 2. to determine the necessity for routine cardiological and respiratory screening.

Study design: This is an observational study. A standard medical history, neurological examination, functional measures, questionnaires, cardiac examination, respiratory function tests, radiological examination (qualitative and quantitative full body MRI, muscle ultrasound, DEXA scan, X-ray of the spine) and accelerometry will be performed. For each participant, the investigators will perform four six-monthly measurements over an one-and-a-half year period. If more than 20 patients are willing to participate in this study, the investigators will select per muscle disease 10 participants that are representative of the entire patient population (based on age, gender, disease severity etc.). Patients that are not included in this study and patients that are not able to or do not wish to visit the Radboudumc will be retrospectively analyzed through medical records. Additionally, they will receive questionnaires, which can be completed at home.

Study population: all patients with congenital myopathy/muscular dystrophy due to mutations in the SELENON or LAMA2 genes.

Risk and benefit assessment: This study does not concern any product (medicinal product, food product, or medical device). There is a small risk for minor injury, e.g. when a participant falls. However, since the investigators use all functional test using movements to which most participants are familiar (i.e. walking, transfers, etc), the participant will be able to estimate his/her own risk. The investigators don't include tests in which they push participants to their physical limits. The investigators conclude that this study has a negligible risk. A benefit includes the possibility for participants to get a detailed analysis on their own health. Additionally, participants will contribute to the design of future clinical trials on possible treatment options.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to complete (part of the) measurement protocol
* Willing and able to travel to Nijmegen (The Netherlands)
* Dutch-speaking
* Genetically-confirmed muscle disease caused by mutations in SELENON (SEPN1): congenital muscular dystrophy with early spine rigidity or congenital myopathy (multicore/minicore disease, congenital fiber type size disproportion)
* Genetically confirmed muscular dystrophy caused by mutations in LAMA2: merosin-deficient muscular dystrophy 1A (early-onset LAMA2-related muscular dystrophy) or childhood-onset limb-girdle type muscular dystrophy (late-onset LAMA2-related muscular dystrophy)

Exclusion Criteria:

* None

Ages: 1 Day to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a congenital myopathy/muscular dystrophy due to mutations in SELENON- or LAMA2 genes will be identified through contact with genetic diagnostic services, rehabilitation centers, and muscle disease experts in The Netherlands and Dutch-speaking Belgium. Patients with a congenital myopathy/muscular dystrophy due to SELENON (prevalence 0.5:1000,000) or LAMA2 (4 in 500,000) mutations are rare and no Dutch registry exists. Therefore the investigators can only estimate the number of patients.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2020-08-26 (Actual); Primary Completion 2022-05-23 (Actual); Study Completion 2023-03-24 (Actual)

PRIMARY OUTCOMES:
Change of Motor Function Measure (MFM)-32 (older than 7 years) or MFM-20 (2 to 7 years old) | Change from baseline at 6 months, 12 months and 18 months
  Global motor functioning. The items of the MFM are classified in 3 domains: D1: Standing and transfers (13 items, sub score range 0-39) D2: Axial and proximal motor function (12 items, sub score range 0-36) D3: Distal motor function (7 items, sub score range 0-21) Each item is scored on a 0-3 scale. Each sub score will be calculated as the percentage of total possible score achieved. Higher scores indicate a better outcome. The range of the total score is 0-96, again recalculated as the percentage of total possible score achieved. The main point of interest includes the change of MFM score over a period of 1,5 year. Additionally, MFM scores of participants will be compared to reference values.

SECONDARY OUTCOMES:
Accelerometry (2 years and older) - change of physical activity in daily life | Change from baseline at 6 months, 12 months and 18 months
  Physical activity in daily life will be assessed by wearing an accelerometer (GENEActiv original devices) for 7 days. The main point of interest includes the change of physical activity in daily life over a period of 1,5 year
Change of activity limitations - ACTIVLIM (6 years and older) | Change from baseline at 6 months, 12 months and 18 months
  ACTIVLIM assesses the ability to perform 22 activities of daily life on a 3-point scale from impossible to easy. The main point of interest includes the change of activity limitations over a period of 1,5 year. Additionally, the ACTIVLIM scores of participants will be compared to reference values.
Change of balance by Pediatric balance scale (2 - 17 years) or Mini Balance Evaluation System Test (miniBEST) (18 years and older) | Change from baseline at 6 months, 12 months and 18 months
  Balance will be assessed through the Pediatric balance scale (2 - 17 years) or the Mini Balance Evaluation System Test (miniBEST) (18 years and older). The Pediatric Balance Scale is a modified version of the Berg Balance Scale that is used to assess functional balance skills in school-aged children with mild to moderate motor impairments. The miniBEST evaluates balance control by scoring of exercises that belong to one of the following categories: anticipatory postural changes, reactive postural control, sensory orientation and walking. The main point of interest includes the change of balance scores over a period of 1,5 year. Additionally, the balance score of participants will be compared to reference values.
Change of bone density - DEXA scan (2 years and older) | Change from baseline at 12 months
  The bone density of the spine and hip will be measured by a DEXA scan. The main point of interest includes the change of bone density over a period of 1 year. Additionally, bone density of participants will be compared to reference values.
Change of Borg Rating Scale of Perceived Exertion (5 years and older) - physical activity intensity level | Change from baseline at 6 months, 12 months and 18 months
  Borg Rating Scale of Perceived Exertion is a way of measuring physical activity intensity level. Perceived exertion is based on the physical sensations a person experiences during physical activity. Participants will be asked to score the intensity level at the beginning and at the end of the 6MWT. The main point of interest includes the change of perceived exertion over a period of 1,5 year.
Change of cardiac function (2 years and older) | Change from baseline at 12 months
  Cardiac function will be assessed using standardized cardiac ultrasound protocols with speckle tracking, including global longitudinal strain (GLS), 3D left ventricle ejection fraction (LVEF), right ventricle s' and right ventricle fractional area change (RV FAC) combined with standard electrocardiography (ECG). The main point of interest includes the change of cardiac function over a period of 1 year. Additionally, cardiac function of participants will be compared to reference values.
Change of The Children's Hospital of Philadelphia Infant Test of Neuromuscular Disorders (CHOP INTEND) score (children under the age of 2 years) | Change from baseline at 6 months, 12 months and 18 months
  CHOP INTEND has been shown to be valid for the assessment of motor skills of children below 2 years of age. The main point of interest includes the change of CHOP INTEND score over a period of 1,5 year. Additionally, the CHOP INTEND score of participant will be compared to reference values.
Change of fatigue (adults, 18 years and older) - Checklist Individual Strength (CIS) | Change from baseline at 6 months, 12 months and 18 months
  The CIS is a questionnaire rating four subscales: subjective tiredness, concentration, motivation and physical activity. It consists of 20 items on a 7-point scale. The main point of interest includes the change of fatigue over a period of 1,5 year. Additionally, fatigue scores of participants will be compared to reference values.
Change of fatigue (pediatric, 2-17 years old) - PedsQL Multidimensional Fatigue Scale (MFS) | Change from baseline at 6 months, 12 months and 18 months
  The PedsQL MFS assesses subjective fatigue in three domains, namely General Fatigue Scale, Sleep/Rest Fatigue Scale, and Cognitive Fatigue Scale. The main point of interest includes the change of fatigue over a period of 1,5 year. Additionally, fatigue scores of participants will be compared to reference values.
Change of functional ability in daily life - Egen klassifikation scale version 2 (EK2) (16 years and older) | Change from baseline at 6 months, 12 months and 18 months
  The EK2 is a questionnaire that was designed to measure functional ability of activities in daily living in non-ambulant Duchenne muscular dystrophy patients. This questionnaire is only available in English. Therefore, only participants of 16 years and older who have a sufficient understanding of the English language will be asked to complete this questionnaire. The main point of interest includes the change of functional ability in daily life over a period of 1,5 year. Additionally, EK2 scores of participants will be compared to reference values.
Change of Functional Ambulation Category (FAC) (5 years and older) | Change from baseline at 6 months, 12 months and 18 months
  The FAC assesses functional ambulation in participants.The main point of interest includes the change of FAC over a period of 1,5 year.
Change of Graded and Timed function tests | Change from baseline at 6 months, 12 months and 18 months
  The time it takes to complete functions of the lower extremity will be assessed with the 30 seconds sit to stand test, Timed up and Go, and the time it takes to climb 4 stairs and to rise from the floor (2 years and older); 6 minute walking test and 10 meter walking test (5 years and older); The main point of interest includes the change of Graded and Timed function tests over a period of 1,5 year. Additionally, values of the Graded and Timed function tests of participants will be compared to reference values.
Change of Hammersmith Infant Neurological Examination (HINE) (under the age of 2 years) | Change from baseline at 6 months, 12 months and 18 months
  HINE is designed to be a simple and scorable method for evaluating infants from 2 months to 2 years of age. It includes 3 sections that assess different aspects of neurologic function, including neurological examination, developmental milestones and behavioral assessment. The main point of interest includes the change of HINE score over a period of 1,5 year. Additionally, HINE scores of participants will be compared to reference values.
Change of Hammersmith Functional Motor Scale (HFMS) (2 years and older, non-ambulant) | Change from baseline at 6 months, 12 months and 18 months
  The HFMS was originally developed to assess the physical abilities of children with non-ambulant Spinal Muscular Atrophy (SMA). It consists of 20 items that were considered as important to measure the physical functioning of those patients. The main point of interest includes the change of HFMS scores. Additionally, HFMS scores of participants will be compared to reference values.
Change of Impact on Participation and Autonomy (IPA) (18 years and older) | Change from baseline at 6 months, 12 months and 18 months
  Questionnaire about participation and autonomy in daily life. The main point of interest includes the change of IPA scores over a period of 1,5 year. Additionally, IPA scores of participants will be compared to reference values.
Change of maximal voluntary isometric contraction (5 years and older) (Newton) | Change from baseline at 6 months, 12 months and 18 months
  Maximal voluntary isometric contraction will be measured by hand-held dynamometry (both hands, m. biceps brachii, m. quadriceps). The main point of interest includes the change of maximal voluntary isometric contraction over a period of 1,5 year. Additionally, maximal voluntary isometric contraction of participants will be compared to reference values.
McGill pain questionnaire (12 years and older) - Change of location, level and characteristics of pain | Change from baseline at 6 months, 12 months and 18 months
  Questionnaire in which the location, level and characteristics of pain are assessed. The main point of interest is the change of location, level and characteristics of pain over a period of 1,5 year.
Change of muscle atrophy (cm) and fattening (echo-intensity) by muscle ultrasound | Change from baseline at 6 months, 12 months and 18 months
  Muscle atrophy and fattening of the leg, arm, back and abdominal muscles will be assessed by muscle ultrasound.The main point of interest includes the change of muscle atrophy and fattening over a period of 1,5 year. Additionally, muscle atrophy and fattening of participants will be compared to reference values.
Change of muscle fattening, atrophy, inflammation and fibrosis by qualitative and quantitative full body muscle MRI | Change from baseline at 12 months
  A full body muscle MRI will be performed in participants who are able to lie supine and still for 60 minutes (participants of 10 years and older) and who are not dependent on respiratory equipment. Muscle fattening will be assessed by Regions of Interest (ROIs) (quantitative) and modified Mercuri score (semi-quantitative). Atrophy will be assessed by muscle volume score (semi-quantitative). Inflammation will be assessed by Malattia score (semi-quantitative). The presence and pattern of muscle fibrosis will be noted.The main point of interest includes the change of muscle fattening, atrophy, inflammation and fibrosis over a period of 1 year. Additionally, these values will be compared to reference values.
Change of muscle power by muscle power measurements (Medical Research Council (MRC) scale) (2 years and older) | Change from baseline at 6 months, 12 months and 18 months
  Muscle power of individual muscle groups can be assessed by muscle power measurements and graded in correspondence with the MRC scale. The main point of interest includes the change of MRC score in participants over a period of 1,5 year.
Pulmonary function (5 years and older) - change of forced vital capacity (percentage predicted) | Change from baseline at 6 months, 12 months and 18 months
  Obtained with handheld spirometry in sit and supine. The main point of interest includes the change of forced vital capacity over a period of 1,5 year. Additionally, forced vital capacity of participants will be compared to reference values.
Pulmonary function (5 years and older) - change of forced expiratory volume in the first second (liter) (percentage predicted) | Change from baseline at 6 months, 12 months and 18 months
  Obtained with handheld spirometry in sit and supine. The main point of interest includes the change of forced expiratory volume in the first second over a period of 1,5 year. Additionally, change of forced expiratory volume in the first second of participants will be compared to reference values.
Pulmonary function (5 years and older) - change of peak expiratory flow (liter per second) | Change from baseline at 6 months, 12 months and 18 months
  Obtained with handheld spirometry in sit and supine. The main point of interest includes the change of peak expiratory flow over a period of 1,5 year. Additionally, peak expiratory flow in participants will be compared to reference values.
Pulmonary function (5 years and older) - change of vital capacity (percentage predicted) | Change from baseline at 6 months, 12 months and 18 months
  Obtained with handheld spirometry in sit and supine. The main point of interest includes the change of vital capacity over a period of 1,5 year. Additionally, vital capacity in participants will be compared to reference values.
Pulmonary function (5 years and older) - change of peak cough flow (liter per second) | Change from baseline at 6 months, 12 months and 18 months
  Obtained with handheld spirometry in sit. The main point of interest includes the change of peak cough flow over a period of 1,5 year. Additionally, peak cough flow in participants will be compared to reference values.
Pulmonary function (5 years and older) - change of maximal expiratory pressure (cmH2O) | Change from baseline at 6 months, 12 months and 18 months
  Obtained with handheld device. The main point of interest includes the change of maximal expiratory pressure over a period of 1,5 year. Additionally, maximal expiratory pressure of participants will be compared to reference values.
Pulmonary function (5 years and older) - change of maximal inspiratory pressure (cmH2O) | Change from baseline at 6 months, 12 months and 18 months
  Obtained with handheld device. The main point of interest includes the change of maximal inspiratory pressure over a period of 1,5 year. Additionally, maximal inspiratory pressure of participants will be compared to reference values.
Pulmonary function (5 years and older) - change of sniff nasal inspiratory pressure (cmH2O) | Change from baseline at 6 months, 12 months and 18 months
  Obtained with handheld device. The main point of interest includes the change of sniff nasal inspiratory pressure over a period of 1,5 year. Additionally, sniff nasal inspiratory pressure of participants will be compared to reference values.
Pulmonary function - change of diaphragm thickness (mm) | Change from baseline at 6 months, 12 months and 18 months
  Obtained with ultrasound. The main point of interest includes the change of diaphragm thickness over a period of 1,5 year. Additionally, the diaphragm thickness of participants will be compared to reference values.
Pulmonary function - change of diaphragm thickening (ratio) | Change from baseline at 6 months, 12 months and 18 months
  Obtained with ultrasound. The main point of interest includes the change of diaphragm thickening over a period of 1,5 year. Additionally, diaphragm thickening of participants will be compared to reference values.
Pulmonary function - change of diaphragm excursion (cm) | Change from baseline at 6 months, 12 months and 18 months
  Obtained with ultrasound. The main point of interest includes the change of diaphragm excursion over a period of 1,5 year. Additionally, diaphragm excursion will be compared to reference values.
Change of Quality of life (adult, 18 years and older) by SF36/RAND36 | Change from baseline at 6 months, 12 months and 18 months
  The adult Quality of Life is measured by the SF36/RAND36 questionnaire. The SF36/RAND36 addresses eight concepts: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. It also includes a single item that provides an indication of perceived change in health. The main point of interest includes the change of Quality of Life over a period of 1,5 year. Additionally, Quality of Life of participants will be compared to reference values.
Change of Quality of life (adult, 18 years and older) by Individualized Neuromuscular Quality of Life (INQoL). | Change from baseline at 6 months, 12 months and 18 months
  The adult Quality of Life is measured by the Individualized Neuromuscular Quality of Life (INQoL) questionnaire. The INQoL is a validated muscle disease specific measure of quality of life, which can be used for individuals or large samples. The main point of interest includes the change of Quality of Life over a period of 1,5 year. Additionally, Quality of Life of participants will be compared to reference values.
Change of Quality of Life (pediatric, 2-17 years old) by PedsQL generic quality of life | Change from baseline at 6 months, 12 months and 18 months
  The pediatric Quality of Life is measured by PedsQL generic quality of life. The PedsQL generic quality of life questionnaire consists of 8 items on physical functioning, 5 items on emotional functioning, 5 items on social functioning, and 5 items on school functioning. Each item is scored on a 0-4 scale. The items are reversed scored and linearly transformed to a 0-100 scale, so that higher scores indicate a better outcome. The main point of interest includes the change of Quality of Life over a period of 1,5 year. Additionally, Quality of Life of participants will be compared to reference values.
Change of Quality of Life (pediatric, 2-17 years old) by PedsQL neuromuscular module (NMM) | Change from baseline at 6 months, 12 months and 18 months
  The PedsQL NMM questionnaire consists of 25 questions in three domains: Neuromuscular disease, communication and family resources. The main point of interest includes the change of Quality of Life over a period of 1,5 year. Additionally, Quality of Life of participants will be compared to reference values.
Change of range of motion of ankles and elbows | Change from baseline at 6 months, 12 months and 18 months
  The range of motion of the ankles and elbows is noted bilaterally by goniometry. The main point of interest includes the change of range of motion of ankles and elbows over a period of 1,5 year. Additionally, the range of motion of ankles and elbows will be compared to reference values.
Change of spine deformity (degree) (2 years and older) | Change from baseline at 12 months
  Spine deformity (scoliosis, lordosis, kyphosis) will be assessed by a full spine X-ray in lateral and anteroposterior direction in a sitting position and in flexion-extension in a lying position. The main point of interest includes the change of spine deformity over a period of 1 year. Additionally, spine deformity of participants will be compared to reference values.
Change of Brooke and Vignos scale (2 years and older) | Change from baseline at 6 months, 12 months and 18 months
  The Brooke and Vignos scales provide ordinal data to assess the upper and lower extremity functions. The main point of interest includes the change of Brooke and Vignos scale over a period of 1,5 year.
Change of Wong-Baker Faces Pain Scale (2 years and older) | Change from baseline at 6 months, 12 months and 18 months
  The Wong-Baker Faces Pain Scale was originally created for children to help them communicate about their pain. The main point of interest includes the change of the Wong-Baker Faces Pain Scale over a period of 1,5 year.

CONTACTS AND LOCATIONS:
Overall Officials: Nicol Voermans, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboudumc, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
Research data is open access shared upon publication, provided that this complies with privacy regulations. The Donders Repository is the default repository for sharing the investigators' data.

REFERENCES:
- [Background] Witting N, Werlauff U, Duno M, Vissing J. Phenotypes, genotypes, and prevalence of congenital myopathies older than 5 years in Denmark. Neurol Genet. 2017 Mar 21;3(2):e140. doi: 10.1212/NXG.0000000000000140. eCollection 2017 Apr. PMID 28357410
- [Background] Scoto M, Cirak S, Mein R, Feng L, Manzur AY, Robb S, Childs AM, Quinlivan RM, Roper H, Jones DH, Longman C, Chow G, Pane M, Main M, Hanna MG, Bushby K, Sewry C, Abbs S, Mercuri E, Muntoni F. SEPN1-related myopathies: clinical course in a large cohort of patients. Neurology. 2011 Jun 14;76(24):2073-8. doi: 10.1212/WNL.0b013e31821f467c. PMID 21670436
- [Background] Schara U, Kress W, Bonnemann CG, Breitbach-Faller N, Korenke CG, Schreiber G, Stoetter M, Ferreiro A, von der Hagen M. The phenotype and long-term follow-up in 11 patients with juvenile selenoprotein N1-related myopathy. Eur J Paediatr Neurol. 2008 May;12(3):224-30. doi: 10.1016/j.ejpn.2007.08.011. Epub 2007 Oct 22. PMID 17951086
- [Background] Oliveira J, Gruber A, Cardoso M, Taipa R, Fineza I, Goncalves A, Laner A, Winder TL, Schroeder J, Rath J, Oliveira ME, Vieira E, Sousa AP, Vieira JP, Lourenco T, Almendra L, Negrao L, Santos M, Melo-Pires M, Coelho T, den Dunnen JT, Santos R, Sousa M. LAMA2 gene mutation update: Toward a more comprehensive picture of the laminin-alpha2 variome and its related phenotypes. Hum Mutat. 2018 Oct;39(10):1314-1337. doi: 10.1002/humu.23599. Epub 2018 Aug 10. PMID 30055037
- [Background] Nguyen Q, Lim KRQ, Yokota T. Current understanding and treatment of cardiac and skeletal muscle pathology in laminin-alpha2 chain-deficient congenital muscular dystrophy. Appl Clin Genet. 2019 Jul 3;12:113-130. doi: 10.2147/TACG.S187481. eCollection 2019. PMID 31308722
- [Background] Moulin M, Ferreiro A. Muscle redox disturbances and oxidative stress as pathomechanisms and therapeutic targets in early-onset myopathies. Semin Cell Dev Biol. 2017 Apr;64:213-223. doi: 10.1016/j.semcdb.2016.08.003. Epub 2016 Aug 12. PMID 27531051
- [Background] de Vries PR, Janssen M, Spaans E, de Groot I, Janssen A, Smeitink J, Koene S. Natural variability of daily physical activity measured by accelerometry in children with a mitochondrial disease. Mitochondrion. 2019 Jul;47:30-37. doi: 10.1016/j.mito.2019.04.005. Epub 2019 Apr 20. PMID 31014978
- [Derived] Bouman K, van Doorn JLM, Groothuis JT, Wijkstra PJ, van Engelen BGM, Erasmus CE, Doorduin J, Voermans NC. Respiratory function in LAMA2-related muscular dystrophy and SELENON-related congenital myopathy, a 1.5-year natural history study. Eur J Paediatr Neurol. 2024 Jan;48:30-39. doi: 10.1016/j.ejpn.2023.11.005. Epub 2023 Nov 22. PMID 38008001
- [Derived] Bouman K, Groothuis JT, Doorduin J, van Alfen N, Udink Ten Cate FEA, van den Heuvel FMA, Nijveldt R, Kamsteeg EJ, Dittrich ATM, Draaisma JMT, Janssen MCH, van Engelen BGM, Erasmus CE, Voermans NC. LAMA2-Related Muscular Dystrophy Across the Life Span: A Cross-sectional Study. Neurol Genet. 2023 Jul 19;9(5):e200089. doi: 10.1212/NXG.0000000000200089. eCollection 2023 Oct. PMID 37476021
- [Derived] Bouman K, Groothuis JT, Doorduin J, van Alfen N, Udink Ten Cate FEA, van den Heuvel FMA, Nijveldt R, van Tilburg WCM, Buckens SCFM, Dittrich ATM, Draaisma JMT, Janssen MCH, Kamsteeg EJ, van Kleef ESB, Koene S, Smeitink JAM, Kusters B, van Tienen FHJ, Smeets HJM, van Engelen BGM, Erasmus CE, Voermans NC. Natural history, outcome measures and trial readiness in LAMA2-related muscular dystrophy and SELENON-related myopathy in children and adults: protocol of the LAST STRONG study. BMC Neurol. 2021 Aug 12;21(1):313. doi: 10.1186/s12883-021-02336-z. PMID 34384384

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-08): https://cdn.clinicaltrials.gov/large-docs/81/NCT04478981/Prot_SAP_000.pdf